CLINICAL TRIAL: NCT00710346
Title: Establishment of a Fibroid Tissue Bank
Brief Title: Establishment of Fibroid Tissue Bank
Status: Terminated | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080170; 08-CH-0170
Record Dates: First submitted 2008-07-03; First posted 2008-07-04 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2016-09-01

CONDITIONS: Leiomyoma; Fibroids
Keywords: Leiomyoma; Uterus; Fibroids; Surgical
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to collect information and tissue samples from women with uterine fibroids. The samples will be used to study genes, proteins and other substances in order to better understand the disease process and improve fertility and reproductive health.

Women who are scheduled to undergo hysterectomy, myomectomy or other surgery due to uterine fibroids or to an unusual variant of fibroid disease, such as HLRCC or benign metastasizing leiomyomatosis, may be eligible for this study.

Tissue samples are collected from participants during surgery. The samples are coded and catalogued for research use. Data collected regarding the surgery include the sample location, surgery type, reason for surgery and the primary and secondary diagnoses. Additional data collected about the participant include date of birth, race, ethnicity, weight, height, smoking status, information about menstrual cycles, medications and family history.

DETAILED DESCRIPTION:
The long term goal of this protocol is to create a repository of well-characterized fibroid (leiomyoma) tissues in order to gather information that will lead to improved understanding of uterine fibroid growth and pathogenesis. It is expected that this initiative will eventually improve fertility and reproductive health of the millions of women who suffer from fibroids.

To address the need for increased research in this field, the NICHD in collaboration with the Office of Research on Women s Health (ORWH) will establish a national fibroid tissue bank. This initiative will strengthen the science base, improve our understanding of how uterine fibroids develop and grow, and provide clues to more effective conservative management of fibroids. The rationale for this protocol is that a repository of well-characterized, well-preserved leiomyoma tissues will provide investigators interested in basic and translational research on fibroids the opportunity to study the condition. This will facilitate research because experiments conducted on the samples may be expected to improve understanding of the mechanism and pathophysiology of this disease.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Women aged 21-80 with uterine fibroids
* Medically indicated hysterectomy, myomectomy or other surgery for uterine fibroids.
* Samples from patients with unusual variants of fibroid disease (HLRCC, benign metastasizing leiomyomatosis) will be included. These samples may possibly not arise from the uterus proper, as the leiomyoma may have become located elsewhere in the body.

EXCLUSION CRITERIA:

* Inability to give consent or understand the consent forms.
* HIV-infected tissues will be excluded due to concern of equipment contamination.
* Hepatitis-infected tissues will be excluded due to concern of equipment contamination.

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2008-06-30; Study Completion 2016-09-01

CONTACTS AND LOCATIONS:
Overall Officials: Alan H DeCherney, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Marshall LM, Spiegelman D, Barbieri RL, Goldman MB, Manson JE, Colditz GA, Willett WC, Hunter DJ. Variation in the incidence of uterine leiomyoma among premenopausal women by age and race. Obstet Gynecol. 1997 Dec;90(6):967-73. doi: 10.1016/s0029-7844(97)00534-6. PMID 9397113
- [Background] Lepine LA, Hillis SD, Marchbanks PA, Koonin LM, Morrow B, Kieke BA, Wilcox LS. Hysterectomy surveillance--United States, 1980-1993. MMWR CDC Surveill Summ. 1997 Aug 8;46(4):1-15. PMID 9259214
- [Background] Payson M, Leppert P, Segars J. Epidemiology of myomas. Obstet Gynecol Clin North Am. 2006 Mar;33(1):1-11. doi: 10.1016/j.ogc.2005.12.004. PMID 16504803